CLINICAL TRIAL: NCT05996263
Title: Prognostic Value of Combined Approach Based on KEAP1/NFE2L2 Mutations and Pre-therapeutic FDG-PET/CT Radiomic Analysis in Advanced Non-small-cell Lung Cancer PDL1 ≥ 50% Treated With Pembrolizumab.
Brief Title: Prognostic Value of Combined Approach Based on KEAP1/NFE2L2 Mutations and Pre-therapeutic FDG-PET/CT Radiomic Analysis in Advanced Non-small-cell Lung Cancer PDL1 ≥ 50% Treated With Pembrolizumab (PEMBROMIC)
Acronym: PEMBROMIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0142 - PEMBROMIC
Record Dates: First submitted 2023-08-01; First posted 2023-08-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2023-08

CONDITIONS: Lung Cancer Stage III; Lung Cancer Stage IV
Keywords: PDL1; PET/CT; Pembrolizumab; KEAP1/NFE2L2
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pembrolizumab has been approved for first-line locally advanced or metastatic NSCLC with a tumor proportion score (TPS) ≥50% for PDL1, based on the results of KEYNOTE-024.

However, even with a positive PDL1 status, only a fraction of patients respond to immunotherapy. In the KEYNOTE-024 study evaluating pembrolizumab versus chemotherapy in first-line advanced NSCLC with PDL1 TPS ≥50%, the response rate in the pembrolizumab arm alone was 45%. NFE2L2 is a transcription factor that directs the expression of free radical defense genes that may interfere with radiation-induced DNA damage. KEAP1 is an adaptor protein that targets NFE2L2 for ubiquitination and proteasomal destruction as part of normal homeostasis. These new biomarkers are of clinical interest, as KEAP1/NFE2L2 mutations predict radiation resistance in patients with localized NSCLC treated with radiotherapy but not surgery. Some data also suggest a role for the KEAP1/NFE2L2 axis in response to immunotherapy.

Establishing a predictive model for the presence of the KEAP1/NFE2L2 mutation would provide a tool for predicting survival (progression-free and overall), even before the patient starts immunotherapy.

DETAILED DESCRIPTION:
Pembrolizumab has been approved for first-line locally advanced or metastatic NSCLC with a tumor proportion score (TPS) ≥50% for PDL1, based on the results of KEYNOTE-024.

However, even with a positive PDL1 status, only a fraction of patients respond to immunotherapy. In the KEYNOTE-024 study evaluating pembrolizumab versus chemotherapy in first-line advanced NSCLC with PDL1 TPS ≥50%, the response rate in the pembrolizumab arm alone was 45%. This result led to the approval of pembrolizumab for first-line advanced NSCLC with PDL1 TPS ≥ 50%, which nevertheless represents only 22% of patients with stage IIIB/IV NSCLC.

Early identification of biomarkers for patients unlikely to benefit from first-line pembrolizumab is therefore a crucial step in selecting suitable candidates.

Furthermore, in cancer, genomic alterations in NFE2L2, KEAP1 and CUL3 result in constitutive activation of NRF2-dependent gene transcription, which promotes cellular resistance to oxidative stress, xenobiotic efflux, proliferation and metabolic reprogramming. Somatic mutations in NFE2L2 and KEAP1 are found in 3.5-15% and 12-17% of NSCLC patients respectively. NFE2L2 is a transcription factor that directs the expression of free radical defense genes that may interfere with radiation-induced DNA damage. KEAP1 is an adaptor protein that targets NFE2L2 for ubiquitination and proteasomal destruction as part of normal homeostasis. These new biomarkers are of clinical interest, as KEAP1/NFE2L2 mutations predict radiation resistance in patients with localized NSCLC treated with radiotherapy but not surgery. Some data also suggest a role for the KEAP1/NFE2L2 axis in response to immunotherapy.

Establishing a predictive model for the presence of the KEAP1/NFE2L2 mutation would provide a tool for predicting survival (progression-free and overall), even before the patient starts immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically or cytologically proven non-small-cell lung cancer (NSCLC)
* Stage IV NSCLC. Stage III NSCLC unresectable and not amenable to radiotherapy
* PD-L1 expression ≥ 50%.
* No previous systemic treatment for NSCLC.
* Patients treated for 1st-line metastatic disease with immunotherapy alone (pembrolizumab)
* No opposition expressed
* Patient affiliated to a social security scheme

Exclusion Criteria:

* PD-L1 expression <50
* Neuroendocrine tumors
* Secondarily metastatic patients
* Previous treatments
* Opposition formulated
* Patient under legal protection (guardianship, curatorship, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated or being treated with immunotherapy alone with pembrolizumab in 1st-line metastatic NSCLC.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free survival (PFS) | through study completion, an average of 1 year
  PFS is defined as the time elapsed between initiation of treatment and tumor progression or death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 1 year
  OS is defined as the time elapsed between initiation of treatment and death, whatever the cause.

OTHER OUTCOMES:
Robustness of the prediction model | through study completion, an average of 1 year
  Robustness will be assessed by comparing predictions obtained from 2 different blind reviewers

CONTACTS AND LOCATIONS:
Overall Officials: Vincent BOURBONNE, MD, PhD, Principal Investigator — Radiation Oncology Department, Brest University Hospital
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement